CLINICAL TRIAL: NCT01236391
Title: Multicenter Phase 2 Study of Bruton's Tyrosine Kinase (Btk) Inhibitor, PCI-32765, in Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: Safety and Efficacy of PCI-32765 in Participants With Relapsed/Refractory Mantle Cell Lymphoma (MCL)
Acronym: PCYC-1104-CA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1104-CA; PCI-32765 (Other: Pharmacyclics)
Record Dates: First submitted 2010-10-18; First posted 2010-11-08 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Mantle Cell Lymphoma
Keywords: Pharmacyclics; Mantle; Mantle Cell; Lymphoma; Non-Hodgkins; Bortezomib; Velcade; Naive; PCYC
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants received PCI-32765 560 mg daily (Experimental): Participants were enrolled and received 560 mg/day dose, stratified into 2 groups based on prior bortezomib exposure.
  Interventions: Drug: PCI-32765

INTERVENTIONS:
Drug: PCI-32765 — 560 mg daily

SUMMARY:
The primary objective of this study was to evaluate the efficacy of ibrutinib in participants with relapsed or refractory MCL.

The secondary objective was to evaluate the safety of a fixed daily dosing regimen (560 mg daily) of PCI-32765 in this population.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, nonrandomized, multicenter, monotherapy study in subjects with histologically documented MCL who have relapsed after ≥ 1 (but not > 5) prior treatment regimens. All subjects meeting eligibility criteria will receive PCI-32765 capsules at a dosage of 560 mg/day once daily for a 28-day cycle until disease progression, unacceptable toxicity, or enrollment in a long-term extension study, whichever occurs earlier.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* ECOG performance status of ≤ 2
* Pathologically confirmed MCL, with documentation of either overexpression of cyclin D1 or t(11;14), and measurable disease on cross sectional imaging that is ≥ 2 cm in the longest diameter and measurable in 2 perpendicular dimensions
* Documented failure to achieve at least partial response (PR) with, or documented disease progression disease after, the most recent treatment regimen
* At least 1, but no more than 5, prior treatment regimens for MCL (Note: Subjects having received ≥2 cycles of prior treatment with bortezomib, either as a single agent or as part of a combination therapy regimen, will be considered to be bortezomib-exposed.)
* Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations)

Major exclusion criteria:

* Prior chemotherapy within 3 weeks, nitrosoureas within 6 weeks, therapeutic anticancer antibodies within 4 weeks, radio- or toxin-immunoconjugates within 10 weeks, radiation therapy within 3 weeks, or major surgery within 2 weeks of first dose of study drug
* Any life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of PCI-32765 capsules, or put the study outcomes at undue risk
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
* Any of the following laboratory abnormalities:

  1. Absolute neutrophil count (ANC) < 750 cells/mm3 (0.75 x 109/L) unless there is documented bone marrow involvement
  2. Platelet count < 50,000 cells/mm3 (50 x 109/L) independent of transfusion support unless there is documented bone marrow involvement
  3. Serum aspartate transaminase (AST/SGOT) or alanine transaminase (ALT/SGPT) ≥ 3.0 x upper limit of normal (ULN)
  4. Creatinine > 2.0 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2011-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darrin Beaupre, MD, PhD, Study Director — Pharmacyclics LLC.
Locations (18):
- United States (9):
  - Stanford University School of Medicine, Stanford, California
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cll Research and Treatment Program, New Hyde Park, New York
  - New York Presbyterian Hospital/Cornell Medical Center, New York, New York
  - The Ohio Sate university, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia School of Medicine Hospital, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Germany (2):
  - Klinikum der Universitat Munchen - Campus Grosshadern, München
  - Universitatsklinikum Ulm, Klinik fur Innere Medizin II, Ulm
- Poland (3):
  - Oddzail Kliniczny Onkologil, Bydgoszcz
  - Malopolskie Centrum Medyczne, Krakow
  - MTZ Clinical Research Sp. z o.o., Warsaw
- United Kingdom (4):
  - Centre for Experimental Cancer Medicine, London
  - Christie Hospital, Manchester
  - Derriford Hospital, Plymouth
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Wang ML, Blum KA, Martin P, Goy A, Auer R, Kahl BS, Jurczak W, Advani RH, Romaguera JE, Williams ME, Barrientos JC, Chmielowska E, Radford J, Stilgenbauer S, Dreyling M, Jedrzejczak WW, Johnson P, Spurgeon SE, Zhang L, Baher L, Cheng M, Lee D, Beaupre DM, Rule S. Long-term follow-up of MCL patients treated with single-agent ibrutinib: updated safety and efficacy results. Blood. 2015 Aug 6;126(6):739-45. doi: 10.1182/blood-2015-03-635326. Epub 2015 Jun 9. PMID 26059948
- [Derived] Marostica E, Sukbuntherng J, Loury D, de Jong J, de Trixhe XW, Vermeulen A, De Nicolao G, O'Brien S, Byrd JC, Advani R, McGreivy J, Poggesi I. Population pharmacokinetic model of ibrutinib, a Bruton tyrosine kinase inhibitor, in patients with B cell malignancies. Cancer Chemother Pharmacol. 2015 Jan;75(1):111-21. doi: 10.1007/s00280-014-2617-3. Epub 2014 Nov 8. PMID 25381051
- [Derived] Wang ML, Rule S, Martin P, Goy A, Auer R, Kahl BS, Jurczak W, Advani RH, Romaguera JE, Williams ME, Barrientos JC, Chmielowska E, Radford J, Stilgenbauer S, Dreyling M, Jedrzejczak WW, Johnson P, Spurgeon SE, Li L, Zhang L, Newberry K, Ou Z, Cheng N, Fang B, McGreivy J, Clow F, Buggy JJ, Chang BY, Beaupre DM, Kunkel LA, Blum KA. Targeting BTK with ibrutinib in relapsed or refractory mantle-cell lymphoma. N Engl J Med. 2013 Aug 8;369(6):507-16. doi: 10.1056/NEJMoa1306220. Epub 2013 Jun 19. PMID 23782157
- See also: www.pharmacyclics.com — http://www.pharmacyclics.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred fifteen subjects were enrolled and 111 subjects received at least 1 dose of ibrutinib and constitute the all treated population and the safety analysis set.
Groups:
- PCI-32765: Participants received 560 mg daily
Period: Overall Study
Arm/Group | PCI-32765
Started | 111 (Participants who received study treatment)
Completed | 95 (Participants who were on treatment or discontinued treatment due to disease progression or death)
Not Completed | 16

BASELINE CHARACTERISTICS:
Population: One hundred fifteen subjects were enrolled and 111 subjects received at least 1 dose of ibrutinib and constitute the all treated population and the safety analysis set.
Arm/Group | PCI-32765
Number analyzed (Participants) | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 85
Region of Enrollment [Number; unit: participants]
  United States | 78
  Poland | 10
  Germany | 3
  United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Response
Description: The primary endpoint of the study was overall response rate (ORR), defined as the proportion of participants who achieved a best overall response of complete response (CR) or partial response (PR), according to the revised International Working Group Criteria for non-Hodgkin's lymphoma (Cheson et al, 2007), as assessed by the investigator. CR is a complete disappearance of all disease, no new lesions, lymph nodes must have regressed and be PET negative, spleen and liver should not be palpable and without nodules, and bone marrow must be negative. PR is a >/= 50% decrease in the sum of the product of diameters of the target lesions, and >/= 50% decrease of splenic and hepatic nodules from baseline, no new lesions and no increase in the size of liver, spleen or non-target lesions.
Time Frame: The median follow-up time on study for all treated participants is 15.3 (range 1.9 - 22.3) months
Population: Participants who received at least 1 dose of PCI-32765 and constitute the all treated population
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Arm/Group | PCI-32765
Number analyzed (Participants) | 111
percentage of participants with response | 67.6 [58.9 to 76.3]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: Number of participants who had experienced at least one treatment emergent AE
Time Frame: From first dose of PCI-32765 to within 30 days of last dose for each participant or until study closure
Measure: Number; unit: participants
Arm/Group | PCI-32765
Number analyzed (Participants) | 111
participants | 111

3. Secondary Outcome: PCI-32765 and Its Metabolite (PCI-45227) AUC0-24h After Repeat Dosing of PCI-32765
Description: Area under the plasma concentration-time curve using data collected at 0, 1, 2, 4, 6-8, and 24 hours post dose (AUC0-24h)
Time Frame: Performed During the First Month of Receiving PCI-32765
Population: PK samples were collected in a subset of participants (n=48) in this trial (n=111). PK parameters reported here reflects those that were PK evaluable from the 48 participants.
Measure: Mean (Standard Deviation); unit: AUC0-24h (ng*h/mL)
Groups:
- PCI-32765 - Day 8; PCI-45227 (Metabolite)- Day 8: PCI-32765: 560 mg daily
Arm/Group | PCI-32765 - Day 8 | PCI-45227 (Metabolite)- Day 8
Number analyzed (Participants) | 43 | 44
AUC0-24h (ng*h/mL) | 953 (705) | 1263 (707)

4. Secondary Outcome: Mean Change From Baseline to Cycle 5 in EORTC QLQ-C30 Global Health Status Score
Description: Mean change from baseline to Cycle 5 in the European Organisation for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) Global Health Status Score according to EORTC QLQ-C30 Scoring Manual (3rd Edition, 2001). For global health status, positive changes indicated better health status or functioning, and negative changes indicated worsening of health status or functioning. Scale scores range from 0 to 100. A change in 5 to 10 points in either direction represents a small change; 10 to 20 points represents a moderate change and greater than 20 points represents a large change.
Time Frame: From Baseline to Cycle 5 (Week 20)
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- EORTC QLQ-C30: Participants received PCI-32765 560 mg daily and completed the EORTC QLQ-C30 questionnaire at Pre-Dose and at Cycle 5
Arm/Group | EORTC QLQ-C30
Number analyzed (Participants) | 69
scores on a scale | 0.6 (22.4)

ADVERSE EVENTS:
Time Frame: From first dose of PCI-32765 to within 30 days of last dose
Arm/Group | PCI-32765
Serious Adverse Events (participants affected / at risk) | 62/111
Other Adverse Events (participants affected / at risk) | 111/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCI-32765 (N=111)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 5
Atrial flutter (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Ileus paralytic (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 3
Non-cardiac chest pain (General disorders) | 2
Chills (General disorders) | 1
Device leakage (General disorders) | 1
General physical health deterioration (General disorders) | 1
Pneumonia (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Anal abscess (Infections and infestations) | 1
Cellulitis orbital (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster ophthalmic (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia klebsiella (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Transient global amnesia (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 2
Renal failure acute (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCI-32765 (N=111)
Neutropenia (Blood and lymphatic system disorders) | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 20
Anaemia (Blood and lymphatic system disorders) | 14
Leukopenia (Blood and lymphatic system disorders) | 7
Leukocytosis (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lymphocytosis (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 7
Sinus tachycardia (Cardiac disorders) | 5
Sinus bradycardia (Cardiac disorders) | 2
Atrioventricular block first degree (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Torsade de pointes (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Hyperacusis (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Lacrimation increased (Eye disorders) | 8
Cataract (Eye disorders) | 6
Conjunctivitis (Eye disorders) | 6
Dry eye (Eye disorders) | 5
Ocular hyperaemia (Eye disorders) | 2
Vision blurred (Eye disorders) | 2
Visual acuity reduced (Eye disorders) | 2
Vitreous floaters (Eye disorders) | 2
Conjunctival haemorrhage (Eye disorders) | 1
Diabetic retinopathy (Eye disorders) | 1
Eye inflammation (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Periorbital oedema (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Scleral haemorrhage (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 55
Nausea (Gastrointestinal disorders) | 34
Constipation (Gastrointestinal disorders) | 28
Vomiting (Gastrointestinal disorders) | 25
Abdominal pain (Gastrointestinal disorders) | 17
Stomatitis (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 12
Abdominal pain upper (Gastrointestinal disorders) | 6
Dry mouth (Gastrointestinal disorders) | 6
Flatulence (Gastrointestinal disorders) | 5
Gastritis (Gastrointestinal disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Oral pain (Gastrointestinal disorders) | 4
Abdominal discomfort (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Epigastric discomfort (Gastrointestinal disorders) | 3
Gingival oedema (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 2
Tongue ulceration (Gastrointestinal disorders) | 2
Barrett's oesophagus (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Lip blister (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Lip ulceration (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Palatal disorder (Gastrointestinal disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Rectal fissure (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 46
Oedema peripheral (General disorders) | 30
Pyrexia (General disorders) | 18
Asthenia (General disorders) | 12
Influenza like illness (General disorders) | 8
Chills (General disorders) | 6
Chest pain (General disorders) | 4
Mucosal inflammation (General disorders) | 4
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 3
Local swelling (General disorders) | 2
Axillary pain (General disorders) | 1
Chest discomfort (General disorders) | 1
Crepitations (General disorders) | 1
Device leakage (General disorders) | 1
Feeling abnormal (General disorders) | 1
Generalised oedema (General disorders) | 1
Gravitational oedema (General disorders) | 1
Induration (General disorders) | 1
Injection site erythema (General disorders) | 1
Injection site extravasation (General disorders) | 1
Injection site haematoma (General disorders) | 1
Injection site pain (General disorders) | 1
Injection site reaction (General disorders) | 1
Malaise (General disorders) | 1
Oedema (General disorders) | 1
Performance status decreased (General disorders) | 1
Xerosis (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1
Seasonal allergy (Immune system disorders) | 3
Hypersensitivity (Immune system disorders) | 2
Allergy to arthropod bite (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 26
Sinusitis (Infections and infestations) | 14
Urinary tract infection (Infections and infestations) | 14
Pneumonia (Infections and infestations) | 10
Nasopharyngitis (Infections and infestations) | 9
Bronchitis (Infections and infestations) | 8
Cellulitis (Infections and infestations) | 8
Folliculitis (Infections and infestations) | 5
Herpes zoster (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 5
Oral herpes (Infections and infestations) | 4
Skin infection (Infections and infestations) | 4
Clostridium difficile colitis (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 3
Lower respiratory tract infection (Infections and infestations) | 3
Paronychia (Infections and infestations) | 3
Staphylococcal infection (Infections and infestations) | 3
Tooth infection (Infections and infestations) | 3
Bacteraemia (Infections and infestations) | 2
Clostridial infection (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 2
Eye infection (Infections and infestations) | 2
Herpes simplex (Infections and infestations) | 2
Infection (Infections and infestations) | 2
Localised infection (Infections and infestations) | 2
Otitis media (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 2
Wound infection (Infections and infestations) | 2
Bronchiolitis (Infections and infestations) | 1
Citrobacter infection (Infections and infestations) | 1
Conjunctivitis infective (Infections and infestations) | 1
Cryptococcosis (Infections and infestations) | 1
Eye infection bacterial (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Genital infection fungal (Infections and infestations) | 1
Haemophilus infection (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Herpes zoster ophthalmic (Infections and infestations) | 1
Histoplasmosis (Infections and infestations) | 1
Implant site infection (Infections and infestations) | 1
Incision site infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Lip infection (Infections and infestations) | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Onychomycosis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Papilloma viral infection (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Rectal abscess (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Urinary tract infection pseudomonal (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 19
Fall (Injury, poisoning and procedural complications) | 8
Laceration (Injury, poisoning and procedural complications) | 3
Excoriation (Injury, poisoning and procedural complications) | 2
Traumatic haematoma (Injury, poisoning and procedural complications) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1
Eye injury (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Open wound (Injury, poisoning and procedural complications) | 1
Post procedural constipation (Injury, poisoning and procedural complications) | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Skin wound (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 6
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Weight decreased (Investigations) | 3
Weight increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 2
Cardiac murmur (Investigations) | 2
Glomerular filtration rate decreased (Investigations) | 2
International normalised ratio increased (Investigations) | 2
Activated partial thromboplastin time prolonged (Investigations) | 1
Aspergillus test positive (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin abnormal (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood immunoglobulin G decreased (Investigations) | 1
Blood iron decreased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Breath sounds abnormal (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Haemophilus test positive (Investigations) | 1
Heart rate irregular (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Macular reflex abnormal (Investigations) | 1
Mean cell volume increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Urine output decreased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 24
Hyperuricaemia (Metabolism and nutrition disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 12
Hypokalaemia (Metabolism and nutrition disorders) | 9
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Enzyme abnormality (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Alcohol intolerance (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 16
Headache (Nervous system disorders) | 12
Peripheral sensory neuropathy (Nervous system disorders) | 6
Paraesthesia (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 3
Amnesia (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Balance disorder (Nervous system disorders) | 1
Dizziness postural (Nervous system disorders) | 1
Head discomfort (Nervous system disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Migraine with aura (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Nystagmus (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Sensory disturbance (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 11
Anxiety (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 6
Agitation (Psychiatric disorders) | 3
Confusional state (Psychiatric disorders) | 3
Abnormal behaviour (Psychiatric disorders) | 1
Euphoric mood (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 5
Renal failure acute (Renal and urinary disorders) | 4
Pollakiuria (Renal and urinary disorders) | 3
Dysuria (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 2
Azotaemia (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Obstructive uropathy (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Haematospermia (Reproductive system and breast disorders) | 2
Oedema genital (Reproductive system and breast disorders) | 2
Breast pain (Reproductive system and breast disorders) | 1
Penile pain (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 20
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 17
Petechiae (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Skin lesion (Skin and subcutaneous tissue disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 6
Ecchymosis (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 5
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 5
Night sweats (Skin and subcutaneous tissue disorders) | 5
Rash macular (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 3
Onychoclasis (Skin and subcutaneous tissue disorders) | 3
Purpura (Skin and subcutaneous tissue disorders) | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 3
Blister (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Sunburn (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 11
Hypotension (Vascular disorders) | 6
Orthostatic hypotension (Vascular disorders) | 2
Blood pressure fluctuation (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No